CLINICAL TRIAL: NCT01332513
Title: An Open Label, Randomised, Repeat Dose Study to Assess the Pharmacokinetic Performance of Five Ezogabine/Retigabine Modified Release (MR) Formulations at Steady State Compared to the Immediate Release (IR) Formulation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114552
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
Keywords: Healthy Volunteers
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- ABFCED sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 milligram (mg) twice daily (BID) dosing of ezogabine modified release (MR) tablet in periods A, B, C, D and E and will receive 200 mg three times daily (TID) dosing of ezogabine immediate release (IR) tablet in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)
- BCADFE sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 mg BID dosing of ezogabine MR in periods A, B, C, D and E and will receive 200 mg TID dosing of ezogabine IR in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)
- CDBEAF sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 mg BID dosing of ezogabine MR in periods A, B, C, D and E and will receive 200 mg TID dosing of ezogabine IR in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)
- DECFBA sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 mg BID dosing of ezogabine MR in periods A, B, C, D and E and will receive 200 mg TID dosing of ezogabine IR in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)
- EFDACB sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 mg BID dosing of ezogabine MR in periods A, B, C, D and E and will receive 200 mg TID dosing of ezogabine IR in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)
- FAEBDC sequence (Experimental): Each subject will participate in six study periods in the bioavailability phase, wherein the subjects will receive a 300 mg BID dosing of ezogabine MR in periods A, B, C, D and E and will receive 200 mg TID dosing of ezogabine IR in period F. Following the completion of the crossover phase, subjects will be re-randomized to one of five cohorts receiving 600 mg doses of either G, H, I, J or K for the food effect phase.
  Interventions: Drug: Investigational Medicinal Product (MR1); Drug: Investigational Medicinal Product (MR2); Drug: Investigational Medicinal Product (MR3); Drug: Investigational Medicinal Product (MR4); Drug: Investigational Medicinal Product (MR5); Drug: Investigational Medicinal Product (IR)

INTERVENTIONS:
Drug: Investigational Medicinal Product (MR1) — Ezogabine MR1 at a dose strength of 300 mg will be orally administered with approximately 250 milliliter (mL) of water to group A subjects during the bioavailability phase. For the food effect phase subjects in group G will be orally administered MR1 tablets at a dose strength of 600 mg.
Drug: Investigational Medicinal Product (MR2) — Ezogabine MR2 at a dose strength of 300 mg will be orally administered to group B subjects with approximately 250 mL of water during the bioavailability phase. For the food effect phase subjects in group H will be orally administered MR2 tablets at a dose strength of 600 mg.
Drug: Investigational Medicinal Product (MR3) — Ezogabine MR3 will be orally administered with approximately 250 mL of water to group C subjects during the bioavailability phase. For the food effect phase subjects in group I will be orally administered MR3 tablets at a dose strength of 600 mg.
Drug: Investigational Medicinal Product (MR4) — Ezogabine MR4 will be orally administered with approximately 250 mL of water to group D subjects during the bioavailability phase. For the food effect phase subjects in group J will be orally administered MR4 tablets at a dose strength of 600 mg.
Drug: Investigational Medicinal Product (MR5) — Ezogabine MR5 will be orally administered with approximately 250 mL of water to group E subjects during the bioavailability phase. For the food effect phase subjects in group K will be orally administered MR5 tablets at a dose strength of 600 mg.
Drug: Investigational Medicinal Product (IR) — Ezogabine IR at dose strengths of 50 mg and 200 mg will be orally administered with approximately 250 mL of water.

SUMMARY:
This is an open-label, single centre, repeat dose, up- titration study in healthy male and female subjects to assess the pharmacokinetic (PK) performance of five prototypes of ezogabine modified release tablet formulations.

The study will consist of a screening period, a treatment phase (consisting of a titration phase, bioavailability phase and food effect phase) and a post-treatment follow-up visit. The study duration from screening to follow up will be approximately 7 weeks. No study procedures will start before informed consent is obtained. Subjects will remain in the clinical unit for the duration of the treatment period (35 days).

Subjects will receive repeat doses of ezogabine for up to 34 days starting at a dose of 100 mg IR TID (300mg TDD) with a standard meal (to be consumed 30 min prior to dosing) for Days 1-3, on days 4-6 subjects will receive 150mg IR TID (450mg TDD). On Day 7 through to the end of the study subjects will receive ezogabine (Mr or IR) at a dose of 600mgTDD.

On Day 7 subjects will enter into a 6-way cross over period to investigate the 5 MR formulations being tested (each at 300mg BID) and the single IR formulation (at 200mg TID). Subjects will receive each formulaition for 4 days and blood samples for pharmacokinetic analysis will be collected up to 24 hours post dose on each 4th day (PK days).

On Day 31 subjects will enter into a food effect phase to investigate the 5 MR formulations being tested (each at 600mg QD). Subjects in this period will have a PK day on Day 33 (following a standard breakfast), and on Day 34 (following a high fat breakfast) to investigate a food effect on the PK profile of ezogabine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician
2. Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined
   * Child-bearing potential and agrees to use one of the contraception methods listed
4. Male subjects must agree to use one of the contraception methods listed
5. Body weight > 50 kg and body mass index (BMI) within the range of 18 - 30kg/m2 (inclusive).
6. Normal or High Normal blood pressure
7. 24hr holter with no clinically significant findings.
8. QTcB or QTcF < 450 msec at screening and pre-dose.
9. Creatinine Clearance within the normal range at screening and pre-dose.
10. Liver function test within normal limits at screening and pre-dose.
11. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subjects who are vegetarian or vegan, or for any other reason be unwilling to consume a high fat meal.
2. The subject has either a previous disease or current medical condition
3. Has made a suicide attempt in the past or, in the investigator's judgment, poses significant suicide risk.
4. Presence of clinically significant proteinuria or hematuria or other clinically significant findings in urinalysis.
5. Subjects with symptoms of urinary dysfunction.
6. Subjects whose ECG shows PR interval is >220 msec, or presence of intraventricular conduction disturbances (complete or incomplete BBB), at screening or prior to dosing.
7. Presence of clinically significant arrhythmias.
8. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
9. Current or chronic liver disease or biliary abnormalities. Medical history positive for biliary signs and symptoms (cholecystectomy is acceptable).
10. History of regular alcohol consumption within 6 months of the study.
11. A positive drug/alcohol screen at screening and / or pre-dose.
12. A positive test for HIV antibody.
13. The subjects smokes more than 10 cigarettes per week.
14. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
15. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
16. Use of prescription or non-prescription drugs.
17. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
18. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
19. Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
20. Lactating females.
21. Unwillingness or inability to follow the procedures outlined in the protocol.
22. Subject is mentally or legally incapacitated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02-10 (Actual); Primary Completion 2011-05-23 (Actual); Study Completion 2011-05-23 (Actual)

PRIMARY OUTCOMES:
Area under the curve from zero to 24 hours at steady-state of ezogabine | Days 10, 14, 18, 22, 26 and 30

SECONDARY OUTCOMES:
Area under the curve of ezogabine from zero to 24 hours at steady-state | Days 33 and 34
Cmax of ezogabine at steady state | Days 10, 14, 18, 22, 26, 30, 33 and 34
Tmax of ezogabine at steady-state | Days 10, 14, 18, 22, 26, 30, 33 and 34
Cmin of ezogabine at steady state | Days 10, 14, 18, 22, 26, 30, 33 and 34
Cmax:Cmin Ratio of ezogabine | Days 10, 14, 18, 22, 26, 30, 33 and 34
Fluctuation Index (FI) of ezogabine | Days 10, 14, 18, 22, 26, 30, 33 and 34

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114552 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114552?search=study&search_terms=114552#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114552 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register